CLINICAL TRIAL: NCT06171932
Title: Comparison Of Efficacy Of Hydrocortisone And Methyl Prednisolone In Acute Severe Asthma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Inayat Ur Rehman, Principal Investigator, University of Karachi
Other Study IDs: Zia ud din university karachi
Record Dates: First submitted 2023-11-24; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Asthma Acute
MeSH Terms: interventions — Methylprednisolone; Hydrocortisone

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HYDROCORTISONE: Group A will comprise of 30 patients will be treated with 200 mg hydrocortisone followed by 3 doses of hydrocortisone 100 mg 6 hours apart for next 24hrs
- METHYLPREDNISOLONE: Group B will be treated with methylprednisolone 125 mg stat
  Interventions: Drug: Methylprednisolone,

INTERVENTIONS:
Drug: Methylprednisolone, — No intervention required
  Other Names: Hydrocortisone
  Groups: METHYLPREDNISOLONE

SUMMARY:
COMPARISON OF EFFICACY OF HYDROCORTISONE AND METHYLPREDNISOLONE IN ACUTE SEVERE ASTHMA

In this study Investigator will compare the efficacy of hydrocortisone and methyl prednisolone in acute severe asthma that will lead to final result and beneficial effects that will help in early resoloution of symptoms and help in preventing recurrence

DETAILED DESCRIPTION:
investigator will compare the efficacy of hydrocortisone v/s methylprednisolone in management of patients presented with acute severe asthma in emergency.

A local study was conducted in 2009, after that there is a big research gap exists at national level although international literature is available on the same but it can not be generalized to our population due to socio, geographic and economic differences so there is dire need to conduct this study this gives a strong rationale to implement in our settings

ELIGIBILITY:
Inclusion Criteria:

* Either Gender (18 to 50 years old)
* Patient presenting to emergency department with acute severe asthma

Exclusion Criteria:

* Patients with critical illness or pregnant females. .Patient treated other than hydrocortisone and methylprednisolone. .Patients not willing to participate in study.
* Life threatening asthma
* Near fatal asthm

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: 60 30 in each group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-26 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-08 (Estimated)

PRIMARY OUTCOMES:
Spirometry | 24 hours
  Above will be check on arrival of patient to Emergency and post Managment
Blood pressures | 24 hours
  Vital signs at initial presentation and post managment will be recorded Blood pressure in mm HG will be recorded
Respiratory rate | 24 hours
  Respiratory rate at arrival and post managment will be considered Respiratory rate in Breaths/min
Heart rate | 24 hours
  Heart rate beats/min will be checked
PEAK EXPIRATORY FLOW RATE | 24 hours
  it wil be checked on arrival and post managment in Peak Expiratory Flow rate (force expiratory volume in 1 second and force vital capacity )will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Inayat ur Rehman, MD ER, Principal Investigator — zia ud din university karachi
Locations (4):
- Pakistan (4):
  - Zia ud din hospital university, Karachi, Sindh
  - Zia ud din university hospital, Karachi, Sindh
  - Zia ud din university hospitals, Karachi, Sindh
  - Zia ud din university, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: Yes
PERFORMA OF PATIENTS AND DATA TAKEN FROM HOSPITAL OF KARACHI WILL BE SHARED AS WELL RESULT OUTCOME WILL BE SHARED IT WILL INCLUDE STUDY PROTOCOL STATS INFORMED CONSENT CLINICAL STUDY REPORT
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 MONTHS
Access Criteria: IPD CRITERIA WILL SHARE WHEN REQUIRED DIRECTLY FROM INVESTIGASTOR

REFERENCES:
- [Result] Aggarwal P, Bhoi S. Comparing the efficacy and safety of two regimens of sequential systemic corticosteroids in the treatment of acute exacerbation of bronchial asthma. J Emerg Trauma Shock. 2010 Jul;3(3):231-7. doi: 10.4103/0974-2700.66522. PMID 20930966
- See also: Comparision — https://journals.lww.com/onlinejets/fulltext/2010/03030/comparing_the_efficacy_and_safety_of_two_regimens.5.aspx

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-11-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT06171932/Prot_SAP_ICF_000.pdf